CLINICAL TRIAL: NCT05504044
Title: To Study the Effects of Co-ingesting Different Forms of Almond, Almond Paste, Fibre, and Almond Phytochemicals With Bread on Postprandial Glucose and Insulin Profiles
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Singapore Institute of Food and Biotechnology Innovation (Other Government)
Collaborators: Glico Asia Pacific Pte Ltd (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: 2019/00701
Record Dates: First submitted 2022-08-15; First posted 2022-08-17 (Actual); Last update posted 2023-08-31 (Actual); Status verified 2022-08

CONDITIONS: Cardiovascular Diseases; Metabolic Disease
Keywords: Nuts
MeSH Terms: conditions — Cardiovascular Diseases; Metabolic Diseases | interventions — Glycemic Control; Inulin

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Control: Glucose (Other): 50 g glucose dissolved in 250 mL water
  Interventions: Other: Glucose control
- Control: Bread (Other): 91.4 g white bread
  Interventions: Other: Bread control
- Bread and Almond paste (Experimental): 88.7 g white bread and 15 g almond paste
  Interventions: Other: Almond paste
- Bread, Almond paste and Inulin (Experimental): 88.7 g white bread, 15 g almond paste and 4 g inulin
  Interventions: Other: Almond paste and inulin
- Bread, Low dose almond paste and Inulin (Experimental): 89.6 g white bread, 10 g almond paste and 3.8 g inulin
  Interventions: Other: Low dose almond paste and inulin

INTERVENTIONS:
Other: Glucose control — 50 g glucose dissolved in 250 mL water
  Arms: Control: Glucose
Other: Bread control — 91.4 g white bread
  Arms: Control: Bread
Other: Almond paste — 88.7 g white bread and 15 g almond paste
  Arms: Bread and Almond paste
Other: Almond paste and inulin — 88.7 g white bread, 15 g almond paste and 4 g inulin
  Arms: Bread, Almond paste and Inulin
Other: Low dose almond paste and inulin — 89.6 g white bread, 10 g almond paste and 3.8 g inulin
  Arms: Bread, Low dose almond paste and Inulin

SUMMARY:
Food is emerging as the new medicine. There has been growing evidence of the beneficial effects of foods, including nuts on human health. Modulation of both glucose and insulin are at the heart of reducing the risk of cardiovascular and other metabolic diseases. The contribution that nuts have on human health has been studied extensively and it is well established that the consumption of nuts revealed improvements in both blood glucose profile and reduced the risk of coronary heart diseases. Nuts, such as almonds, are nutrient-dense foods that are particularly rich in a-tocopherol. They are excellent sources of protein (~25% of energy) and fibre, low in saturated fatty acid content (4-6%) and high in monounsaturated fatty acids. They also contain significant amounts of essential micronutrients such as folate (B vitamin) and polyphenols. Recently, strong interests on the health effects of nuts improving metabolic syndrome and controlling diabetes has been reported. Preliminary studies have indicated that the inclusion of nuts in the diets of individuals with diabetes and/or metabolic syndrome may improve postprandial glycaemic response, and lipid metabolism in the long run.

ELIGIBILITY:
Inclusion Criteria:

* Chinese Males
* Age: 21-60 years
* Body mass index (BMI) between 18 to 25 kg/m2
* Normal blood pressure (< 140/90 mmHg)
* Fasting blood glucose (FBG) </= 6 mmol/L

Exclusion Criteria:

* People who have any major organ dysfunction (eg. cardiovascular, respiratory, hepatic, renal, gastrointestinal) that may influence taste, olfaction, appetite, digestion, metabolism, absorption or elimination of test foods, nutraceutical or drug
* People who smoke
* People with any genetic and/or metabolic diseases (such as diabetes, hypertension etc)
* People who have medical conditions and/or taking medications known to affect glycaemia (glucocorticoids, thyroid hormones, thiazide diuretics)
* People with known glucose-6-phosphate dehydrogenase deficiency (G6PD deficiency)
* People who have any severe food allergy (e.g. anaphylaxis to peanuts) or any known food allergy/intolerance
* People who consume fibre supplements or other supplements that is likely to interfere with study outcomes

  •• People who have active Tuberculosis (TB) or currently receiving treatment for TB
* People who have any known Chronic infection or known to suffer from or have previously suffered from or is a carrier of Hepatitis B Virus (HBV), Hepatitis C Virus (HCV), Human Immunodeficiency Virus (HIV)
* People who is a study team member or an immediate family of any study team member. Immediate family member is defined as a spouse, parent, child, or sibling, whether biological or legally adopted.
* People is enrolled in a concurrent research study judged not to be scientifically or medically compatible with the study of the CNRC.
* People who have intentionally restrict food intake
* People who have poor veins impeding venous access
* People who have any history of severe vasovagal syncope (blackouts or near faints) following blood draws
* People who partake in sports at the competitive and/or endurance levels

Ages: 21 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2019-10-25 (Actual); Primary Completion 2023-01-18 (Actual); Study Completion 2023-01-18 (Actual)

PRIMARY OUTCOMES:
Postprandial glucose response | 0, 15, 30, 45, 60, 90, 120, 150, 180 minutes
Postprandial insulin response | 0, 15, 30, 45, 60, 90, 120, 150, 180 minutes
GI calculation for the composite meal | 0, 15, 30, 45, 60, 90, 120, 150, 180 minutes

SECONDARY OUTCOMES:
Postprandial low-density lipoprotein cholesterol (LDL) level | 0, 15, 30, 45, 60, 90, 120, 150, 180 minutes
Postprandial high-density lipoprotein cholesterol (HDL) level | 0, 15, 30, 45, 60, 90, 120, 150, 180 minutes
Postprandial total cholesterol (TC) level | 0, 15, 30, 45, 60, 90, 120, 150, 180 minutes
Postprandial triglyceride level | 0, 15, 30, 45, 60, 90, 120, 150, 180 minutes

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical Nutrition Research Centre, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bi X, Yeo MTY, Jeyakumar Henry C. Almond paste and dietary fibre: a novel way to improve postprandial glucose and lipid profiles? Int J Food Sci Nutr. 2022 Dec;73(8):1124-1131. doi: 10.1080/09637486.2022.2141207. Epub 2022 Nov 3. PMID 36329602